CLINICAL TRIAL: NCT06117995
Title: Intrauterine Insemination Outcomes Based on WHO 2021 Manual Assessment of Total Rapidly Progressing Motile Sperm Count
Brief Title: Sperm Motility and IUI Live Birth Rate
Acronym: IUI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: Mỹ Đức Phú Nhuận Hospital (Unknown); Phương Chi Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 02/23/DD-BVMD
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-03

CONDITIONS: Infertility
Keywords: sperm motility; rapid progressive motile sperm; WHO 2021; intrauterine insemination; live birth rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile couples have indication of IUI: Infertile couples have an indication of IUI
  Interventions: Other: Assessment the pre-washed sperm motility before IUI

INTERVENTIONS:
Other: Assessment the pre-washed sperm motility before IUI — The pre-washed sperm motility will be assessed by using WHO 2021 guidelines, stratified into four groups.

SUMMARY:
This prospective cohort study aims to establish a cut-off threshold for pre-washed total rapidly motile sperm count (TRMSC) based on WHO 2021 criteria to predict the live birth rate following intrauterine insemination (IUI). The study seeks to answer two key questions:

1. Is there a correlation between TRMSC, as per the WHO 2021 criteria, and the live birth rate after IUI?
2. What is the appropriate cut-off threshold of TRMSC to predict a positive live birth outcome after IUI? Couples undergoing ovulation induction and IUI for indicated reasons will participate in the study. On the day of insemination, the pre-washed semen from the husband will be assessed according to the WHO 2021 criteria. The outcomes of the IUI procedure will be documented.

DETAILED DESCRIPTION:
Eligible patients will be enrolled in the study on the day of intrauterine insemination (IUI). Both spouses will receive detailed information about the study and provide informed consent. Sperm motility will be evaluated according to the WHO 2021 guidelines before filtration and washing.

Ovarian stimulation will be conducted using human menopausal gonadotropins (hMG) with regular ultrasound monitoring of follicular development. Once the lead follicle reaches a size of 18mm, ovulation will be induced using hCG. If six or more follicles reach a size of 14mm, the patient will be advised to cancel the cycle or consider in-vitro fertilization (IVF). IUI will be performed 36-38 hours after hCG injection.

For patients who prefer non-injection-based ovarian stimulation, an oral agent using letrozole will be offered. Letrozole with a dosage of 5 to 7.5 mg will be administered orally from days 2-5 of the menstrual cycle, and ovarian follicle development will be assessed through ultrasound on day 10.

Sperm samples will be collected through masturbation at the hospital after a period of 2-5 days of ejaculation abstinence. Motility analysis will be performed based on the WHO 2021 guidelines, which classify sperm as rapid progressive (A), slow progressive (B), non-progressive (C), or immotile (D), using the formula: percentage of rapid progressive sperm x density x volume. Semen parameters, including volume, density, and normal morphology ratio, will also be evaluated according to the WHO 2021 guidelines.

The collected sample will undergo processing using the density gradient method, following the WHO 2021 guidelines. The processed semen will be used for IUI, and its concentration and motility will be examined.

During the insemination procedure, a Gynétic soft catheter will be used. After the procedure, the patient will rest for 15 - 20 minutes, followed by luteal-phase support using vaginal micronized progesterone for 14 days. The presence of hCG in the blood will be tested after 14 days to determine a biochemical pregnancy. Confirmation of clinical pregnancy will be based on ultrasound observation of a gestational sac at 7 weeks of gestational age. Prenatal care until delivery will be provided either at specified hospitals or through regular contact.

During delivery, data on labour, delivery, and any complications experienced by the participant or newborn will be collected. Participants who cannot attend prenatal care at the designated hospitals will be contacted regularly for data collection. Descriptive analysis will be used to describe the background characteristics of the study population, presenting continuous variables as means and standard deviations (SD) and comparing them using appropriate statistical tests. Categorical variables will be presented as percentages and compared using relevant statistical tests such as Pearson's chi-square or Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing IUI
* Undergone <4 previous IUI cycles
* Total progressive motility sperm count before sperm preparation: > 5million
* Agree to participate in the study

Exclusion Criteria:

* Using frozen semen

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Live babies born in couples undergo intrauterine insemination
Sampling Method: Probability Sample
Enrollment: 536 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | At 24 weeks of gestation
  Live birth is defined as the complete expulsion or extraction from a woman of a product of fertilization, after 24 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 500 grams or more can be used if gestational age is unknown. In the analysis for the primary endpoint, twin delivery will be considered.

SECONDARY OUTCOMES:
Total motile sperm count after sperm preparation | At 5 minutes after sperm preparation for IUI
  Total motile sperm count after sperm preparation, measured by million sperm
Biochemical pregnancy rate | At 14 days after insemination
  Biochemical pregnancy defined as a serum beta-hCG level greater than 25 mIU/ml at day 14 after insemination
Clinical pregnancy rate | At 7 weeks of gestation
  Clinical pregnancy defined as the presence of at least one gestational sac on ultrasound at week 7 of gestation with the detection of heart beat activity, after insemination
Miscarriage rate | Before 22 weeks of gestational age
  Miscarriage defined as spontaneous loss of a clinical pregnancy before week 22 of gestational age, in which the embryo(s) or fetus(es) is/are nonviable and is/are not spontaneously absorbed or expelled from the uterus.
Multiple pregnancy rate | At 7 weeks of gestation
  Multiple pregnancy defined as two or more gestational sacs or two or more positive heart beats by transvaginal sonography
Preterm delivery rate | At birth
  Preterm delivery is defined as any delivery at <24, <28, <32, <37 completed weeks' gestation
Gestational age at delivery | At birth
  Gestational age at delivery.
Birth weigh | At birth
  Weight of newborn
Stillbirth rate | After 28 completed weeks of gestational age
  Stillbirth defined as the death of a fetus prior to the complete expulsion or extraction from its mother
Congenital abnormalities rate | At birth
  Any congenital abnormalities detected in the newborn

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, Principal Investigator — Mỹ Đức Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8421663/
- See also: Related Info — https://link.springer.com/article/10.1186/s40738-020-00092-1
- See also: Related Info — https://link.springer.com/article/10.1007/s43032-020-00408-y
- See also: Related Info — https://link.springer.com/article/10.1007/s10815-014-0306-0